CLINICAL TRIAL: NCT03282331
Title: Lung MORphological Modifications Evaluated by Electrical Impedance Tomography During Preoxygenation for the Intubation of Hypoxemic Patients: Comparison of Standard Oxygenation, High Flow Nasal Oxygen Therapy, and NonInvasive Ventilation (MORPHEIT Study, an Ancillary Study of PREONIV Trial)
Acronym: MORPHEIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CHU-345; 2012-A00778-35 (Other: 2012-A00778-35)
Record Dates: First submitted 2017-09-04; First posted 2017-09-13 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Adult Patients; Requiring Intubation; Hypoxemia (Defined by PaO2/FiO2( Fraction of Inspired Oxygen) Below 200); Patient Covered by French Health Care System
Keywords: Preoxygenation; Intubation; Electrical Impedance Tomography; Lung aeration; Alveolar recruitment
MeSH Terms: conditions — Hypoxia | interventions — Noninvasive Ventilation

STUDY DESIGN:
Masking Description: open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard oxygenation (Experimental): Electrical impedance tomographic evaluation of lung morphology variations according to the preoxygenation technique : Comparison of Standard Oxygenation, High Flow Nasal Oxygen Therapy, and NonInvasive Ventilation
  Interventions: Procedure: Standard oxygenation
- High flow nasal oxygen therapy (Other): Electrical impedance tomographic evaluation of lung morphology variations according to the preoxygenation technique : Comparison of Standard Oxygenation, High Flow Nasal Oxygen Therapy, and NonInvasive Ventilation
  Interventions: Procedure: High flow nasal oxygenation
- NonInvasive Ventilation (Other): Electrical impedance tomographic evaluation of lung morphology variations according to the preoxygenation technique : Comparison of Standard Oxygenation, High Flow Nasal Oxygen Therapy, and NonInvasive Ventilation
  Interventions: Procedure: noninvasive ventilation

INTERVENTIONS:
Procedure: Standard oxygenation — Electrical impedance tomographic evaluation of lung morphology variations according to the preoxygenation technique : Comparison of Standard Oxygenation, High Flow Nasal Oxygen Therapy, and NonInvasive Ventilation
  Arms: standard oxygenation
Procedure: High flow nasal oxygenation — Electrical impedance tomographic evaluation of lung morphology variations according to the preoxygenation technique : Comparison of Standard Oxygenation, High Flow Nasal Oxygen Therapy, and NonInvasive Ventilation
  Arms: High flow nasal oxygen therapy
Procedure: noninvasive ventilation — Electrical impedance tomographic evaluation of lung morphology variations according to the preoxygenation technique : Comparison of Standard Oxygenation, High Flow Nasal Oxygen Therapy, and NonInvasive Ventilation
  Arms: NonInvasive Ventilation

SUMMARY:
Prospective, randomized clinical multicentric study, in ICU, during preoxygenation for the intubation of hypoxemic patients.

Electrical impedance tomographic evaluation of lung morphology variations according to the preoxygenation technique : Comparison of Standard Oxygenation, High Flow Nasal Oxygen Therapy, and NonInvasive Ventilation

DETAILED DESCRIPTION:
Preoxygenation before endotracheal intubation in the ICU is a prerequisite to limit complications, ranging from desaturation, severe hypoxemia and bradycardia with potential cardiac arrest and death. International recommendations suggest the use of non-invasive ventilation (NIV) technique whenever possible. High flow nasal cannula (HFNC) has recently gained growing interest in the ICU as a treatment of acute respiratory failure, to improve extubation success and as a preoxygenation device before endotracheal intubation. Conflicting results have been published.

The PREONIV study was designed to compare NIV, HFNC and conventional preoxygenation with valve bag mask for the preoxygenation before endotracheal intubation.

Investigator propose to add a lung morphology analysis during preoxygenation. Electrical impedance tomography (EIT) is a non invasive tool which analyse lung aeration variations via the evolution of local thoracic impedances with electrical loop circulating around a thoracic belt with electrodes.

The hypothesis is that the technique of preoxygenation might correlate with oxygen desaturation and potential intubation related complications (PREONIV study). Moreover lung morphology modifications evaluated by EIT might be associated with the preoxygenation technique (MORPHEIT study).

Investigator wish to asses lung morphological modifications evaluated by EIT during preoxygenation in a prospective non blinded randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

* • adults patients

  * requiring intubation and hypoxemia (defined by PaO2/FiO2 below 200)
  * patient covered by french health care system
  * patient included in Hopital Estaing, Clermont-Ferrand

Exclusion Criteria:

* • patient refusal

  * intubation for other causes (excluding hypoxemia)
  * impossibility to measure pulse oxymetry value
  * contraindication for NIV : vomiting
  * NIV intolerance
  * cardiac arrest during intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06-02 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
evolution of lung aeration evaluated by electrical impedance tomography during the preoxygenation for intubation of hypoxemic patients and the arterial blood oxygenation | at day 1

SECONDARY OUTCOMES:
electrical impedance tomography related indexes | at day 1 (before, during and after preoxygenation and at 5 minutes and at 30 minutes after intubation)
Lung inhomogeneity index | at day 1 (during and after preoxygenation and at 5 minutes and at 30 minutes after intubation)
End expiratory lung impedance | at day 1 (during and after preoxygenation and at 5 minutes and at 30 minutes after intubation)
Center of Ventilation | at day 1 (during and after preoxygenation and at 5 minutes and at 30 minutes after intubation)
Tidal Volume | at day 1 (during and after preoxygenation and at 5 minutes and at 30 minutes after intubation)
pulse oxymetry value | at day 1 (at 5 minutes and at 30 minutes after intubation)
Partial pressure of arterial oxygen (PaO2) | at day 1
Regurgitation rate | at day 1
oxyhemoglobin desaturation below 80 % | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Thomas GODET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France